CLINICAL TRIAL: NCT05348655
Title: Impact of the Covid-19 Pandemic on the Epidemiology of Respiratory Syncytial Virus in the Metropolis of Lyon
Brief Title: Impact of the Covid-19 on RSV Epidemic in the Metropolis of Lyon
Acronym: IPCoVRS-2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 502_3
Record Dates: First submitted 2022-04-26; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Rhinovirus; RSV Infection in Children Less Than 5 Years of Age
Keywords: RSV epidemic; Covid-19-RSV interaction; Non-pharmacological-interventions; Bronchiolitis; Asthma; Pneumonia
MeSH Terms: conditions — Bronchiolitis; Asthma; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre Covid-19 cohort: Children hospitalized in the Pediatric Department of the " Hôpital Femme Mère Enfant ", Lyon, France with a RT-PCR positive for RSV during the 2019-2020 winter epidemic
  Interventions: Other: epidemiology
- Per Covid-19 cohort: Children hospitalized in the Pediatric Department of the " Hôpital Femme Mère Enfant ", Lyon, France with a RT-PCR positive for RSV during the 2020-2021, 2021-2022, 2022-2023, and 2023-2024 epidemic. The need for continuation of the study will be reassessed after each season
  Interventions: Other: epidemiology

INTERVENTIONS:
Other: epidemiology — To review of medical records to describe diagnosis and severity of the disease
  Other Names: Medical records analysis
Other: epidemiology — To compare pre- and per-Covid-19 epidemics in terms of numbers of admissions, and proportion of severe disease.
  Other Names: Comparison of cohorts

SUMMARY:
The magnitude of seasonal RSV epidemics brings each year new logistical challenges for the hospitalization of young infants with bronchiolitis that overwhelm hospital capacities and lead to specific winter plans with deprogramming and mobilization of human and logistical resources. The Covid-19 pandemic has changed the way winter epidemics are presented. For example, the seasonal RSV epidemic was shifted by several months in Lyon, with an impression of a lower incidence of hospitalized cases, with a population of older children and with fewer signs of clinical severity. This is largely attributable to the widespread use of barrier gestures and social distancing measures, known as "non-pharmacological interventions" or NPI. Given the magnitude of the reduction of the RSV epidemic, it is legitimate to analyze the benefits of NPIs to draw lessons for maintaining preventive measures around RSV-vulnerable populations; moreover, new preventive pharmacological interventions are soon to be marketed, whether they are particularly refined and long half-life anti-RSV monoclonal antibodies, RSV vaccines for mothers or for newborns and infants. In this perspective, it is crucial to properly define the populations at risk of severe disease to establish a legitimate hierarchy in the implementation of different preventive strategies. The study of the RSV epidemic is a high potential model because of the convergence of epidemiological, virological, and pharmacological knowledge. However, the study of the impact of the pandemic on the epidemiology of rhinovirus also seems promising because, for reasons unknown to date, it seems that the pandemic did not have the same reducing impact on the rhinovirus epidemic; in the latter case, the interest is to confirm the resistance of this virus and to look for more fundamental explanations, for example, on viral interactions.

On a previous study (see NTC 04944160), 519 infants were recruited in the Pre-Covid-19 season population, and 277 infants were recruited in the first Per-Covid-19 season population.

ELIGIBILITY:
Inclusion Criteria:

* Child hospitalized at " Hôpital Femme Mère Enfant ", Lyon, France
* Positive RSV-PCR

Exclusion Criteria:

* Parent's refusal to participate

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children hospitalized in the Pediatric Department of the " Hôpital Femme Mère Enfant ", Lyon, France with a RT-PCR positive for RSV
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Annual evolution of the number and severity of RSV-infection in hospitalized children during per-Covid-19 epidemic compared to pre-Covid-19 pandemic. | Day 0
  Description of number of cases for each clinical picture according to pre-SARS-CoV-2 pandemic and per-SARS-CoV-2 pandemic year.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Virology Lab, Lyon
  - Pediatric Departement, Lyon